CLINICAL TRIAL: NCT02161302
Title: THE EFFECT OF TRANSCRANIAL DIRECT CURRENT STIMULATION (tDCS) IN THE TREATMENT OF CHRONIC PELVIC PAIN ASSOCIATED WITH ENDOMETRIOSIS
Brief Title: THE EFFECT OF tDCS IN THE TREATMENT OF CHRONIC PELVIC PAIN ASSOCIATED WITH ENDOMETRIOSIS
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0092
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain; Endometriosis
Keywords: Endometriosis; Transcranial Direct Current Stimulation; tDCS; Near Infrared Spectroscopy; NIRS; Chronic Pelvic Pain
MeSH Terms: conditions — Chronic Pain; Endometriosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active tDCS (Experimental): tDCS will be applied in the head of the patients in 20 minute sessions, daily from Monday to Friday for 2 weeks (10 sessions total). The stimulation will be administered with a pair of surface electrodes, sponge coated, soaked in saline. A battery-powered constant current stimulator will be used for this purpose (tDCS device Soterix 1X1). The stimulation is performed by placing the anodal electrode in the primary motor cortex (M1) and the cathodal one in the contralateral supraorbital area, and it will use a 2 mA current.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- tDCS Sham (Sham Comparator): The sham tDCS consists of the same montage of the active tDCS, but the device is turned off 30 seconds after initiating stimulation (without letting the patient notice it). Rest of the montage is kept identical as the active one during the 20 minutes that the session lasts.
  Interventions: Device: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — The stimulation will be administered with a pair of surface electrodes, sponge coated, soaked in saline. A battery-powered constant current stimulator will be used for this purpose (tDCS device Soterix 1X1). The stimulation is performed by placing the anodal electrode in the primary motor cortex (M1) and the cathodal one in the contralateral supraorbital area and it will use a 2 mA current.
  Other Names: tDCS
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation — The sham tDCS consists of the same montage of the active tDCS, but the device is turned off 30 seconds after initiating stimulation (without letting the patient notice it). Rest of the montage is kept identical as the active one during the 20 minutes that the session lasts.
  Other Names: Sham tDCS
  Arms: tDCS Sham

SUMMARY:
The purpose of this study is to determine if transcranial direct current stimulation (tDCS) is effective in the treatment of chronic pelvic pain associated with endometriosis

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old, non-menopausal, with the diagnosis of endometriosis by videolaparoscopy and biopsy, able to understand and write the Portuguese language, in treatment with isolated progestin for at least one month, who have the worst daily pain in the analogue visual scale > 4 cm on most of the days in the last month

Exclusion Criteria:

* left-handed women, endometriosis implantation in intestine, bladder or urether (surgical treatment indication), history of intense or frequent headache, chronic dermatologic disease, previous adverse effects to treatment with tDCS, seizures, severe cranial trauma with alteration of the cranial anatomy, metallic intracranial implants or pacemaker, history of pelvic inflammatory disease, non-compensated psychiatric disease, non-collaborative patients, history of neurologic, oncologic disease, heart, renal or hepatic failure.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in worst daily pain assessed with the visual analogue scale. | Once Daily. Start 7 days before treatment, everyday during treatment period and every day during follow-up period (total = 35 days)
  Patients will be asked to write down their worst pain level (assessed by the Visual Analogue Scale, self-administered) in a paper diary with different scores: global pain, pain during menses, pain during sexual intercourse, pain during urination, pain during defecation. They will also be asked to daily write the analgesic drug intake. Total evaluations: 35 days.
Changes in motor cortex blood flow assessed by near infrared spectroscopy | Treatment Day 1 (before receiving the 1st session of tDCS); Day 15 (at the end of treatment period) and Day 29 (at the end of follow-up period)
  Motor cortex blood flow will be assessed before the first session of tDCS (on Treatment day 1), after the end of treatment period (Day 15) and after the follow-up period (Day 29). Total = 3 evaluations.
Change in Functional Pain Scale | Once a week - Treatment Day 1, Day 8, Day 15, Day 22, Day 29
  The Functional Pain Scale will be assessed by the Brazilian Profile of Chronic Pain: Screen (B-PCP:S) once a week, as follows: on Treatment Day 1 (before the first session of tDCS, considered baseline), on Treatment Day 8, Day 15, Day 22, and Day 29. Total = 5 evaluations.
Change in the temperature pain threshold | up to Day 29
  It will be assessed by the Quantitative Sensory Test (QST) in the dominant (right) forearm. The heat pain tolerance and pain threshold to the heat and the temperature defined as pain 6/10 by the participant. The temperature starts at 32°C, and it heat at a 1.0 °C/sec rate and cools down after a button is pressed or whenever it reaches the max temperature of 52°C. The participant will be asked to press the button at the first sensation of pain to determine the pain threshold; to press the button whenever she can not stand the heat anymore for the pain tolerance determination and, for last, to press the button at the temperature she fells pain equivalent to 6/10 in the numeric scale of pain. The pain threshold and the temperature of pain 6/10 will be determined by the arithmetic mean of 3 evaluations each. Total of 3 test days: Day 1 (before the first session of tDCS), after the end of the Treatment period (Day 15) and at the end of the follow-up period (Day 29).
Change in effect of the descendent modulator system of pain | up to Day 29
  It will be assessed by the Conditioned Pain Modulation test (CPM). A nociceptive tonic conditioning stimulus - immersion of the non-dominant hand in cold water (0°C for 1 minute) - will be applied concomitant to the progressive thermal stimulus in the dominant forearm as applied in the QST pattern until it reaches the 6/10 pain temperature previously determined by the participant. It will be tested in Treatment Day 1 (before the first session of tDCS - considered baseline), after the end of the Treatment period (Day 15) and at the end of the follow-up period (Day 29) - Total = 3 evaluation.

SECONDARY OUTCOMES:
Change in serum biomarkers level: The brain derived neurotrophic factor (BDNF) and interleukins | up to Day 29
  A blood sample will be collected to measure BDNF and interleukins on Treatment Day 1 (right before the first tDCS session - considered baseline), after the end of the treatment period (day 15,) and after the end of the follow-up period (day 29). Total = 3 evaluations

OTHER OUTCOMES:
Depressive symptoms level | Treatment Day 1 (before receiving the 1st session of tDCS); Day 15 (at the end of treatment period) and Day 29 (at the end of follow-up period)
  Depression symptoms will be assessed by using the Beck II Inventory. It will be assessed before the first session of tDCS (on Treatment day 1), after the end of treatment period (Day 15) and after the follow-up period (Day 29). Total = 3 evaluations.
Anxiety level | Treatment Day 1 (before receiving the 1st session of tDCS); Day 15 (at the end of treatment period) and Day 29 (at the end of follow-up period)
  Anxiety level will be assessed by State-Trait Anxiety Inventory (STAI), adapted to Brazilian Portuguese Language. It will be assessed before the first session of tDCS (on Treatment day 1), after the end of treatment period (Day 15) and after the follow-up period (Day 29). Total = 3 evaluations.
Psychiatric diseases | 1day on patient screening
  Psychiatric diseases will be evaluated by the Structured Clinical Interview for DSM-IV (SCID) in the patient screening. Total = 1 evaluation
Estradiol level | Treatment Day 1 (before receiving the 1st session of tDCS)
  Estradiol blood level will be measured on treatment Day 1 (before receiving the 1st session of tDCS). Total = 1 evaluation
Adverse Effects | up to Day 29
  At the end of each tDCS session, the incidence of any adverse effects - paresthesia, headache, dizziness, nausea, neck pain, burns, redness or pain in the scalp, insomnia, abrupt humor changes and lack of concentration - will be questioned to the participant. Total = 10 evaluations
Pain catastrophizing thoughts | Treatment Day 1 (before receiving the 1st session of tDCS); Day 15 (at the end of treatment period) and Day 29 (at the end of follow-up period)
  The level of catastrophic thinking will be assessed by the Pain Catastrophizing Scale on Treatment Day 1 (before receiving the 1st session of tDCS), after the treatment period (Day 15) and at the end of the follow-up period (Day29). Total = 3 evaluations
Demographic data and comorbidities | Baseline
  Demographic data and comorbidities will be asked in the baseline (before the first session of tDCS). Total = 1 evaluation.
Change in quality of life | Baseline and Day 15
  Quality of life will be assessed by the WHOQOL (World Health Organization Quality of Life), in Treatment Day 1 (before the first session of tDCS - considered baseline) and after the treatment period (Day 15). Total = 2 evaluations

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Valle A, Roizenblatt S, Botte S, Zaghi S, Riberto M, Tufik S, Boggio PS, Fregni F. Efficacy of anodal transcranial direct current stimulation (tDCS) for the treatment of fibromyalgia: results of a randomized, sham-controlled longitudinal clinical trial. J Pain Manag. 2009;2(3):353-361. PMID 21170277
- [Background] Nacul AP, Spritzer PM. [Current aspects on diagnosis and treatment of endometriosis]. Rev Bras Ginecol Obstet. 2010 Jun;32(6):298-307. doi: 10.1590/s0100-72032010000600008. Portuguese. PMID 20945016
- [Background] Boros K, Poreisz C, Munchau A, Paulus W, Nitsche MA. Premotor transcranial direct current stimulation (tDCS) affects primary motor excitability in humans. Eur J Neurosci. 2008 Mar;27(5):1292-300. doi: 10.1111/j.1460-9568.2008.06090.x. Epub 2008 Feb 29. PMID 18312584
- [Background] Nitsche MA, Liebetanz D, Antal A, Lang N, Tergau F, Paulus W. Modulation of cortical excitability by weak direct current stimulation--technical, safety and functional aspects. Suppl Clin Neurophysiol. 2003;56:255-76. doi: 10.1016/s1567-424x(09)70230-2. No abstract available. PMID 14677403
- [Background] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Background] Fenton BW, Palmieri PA, Boggio P, Fanning J, Fregni F. A preliminary study of transcranial direct current stimulation for the treatment of refractory chronic pelvic pain. Brain Stimul. 2009 Apr;2(2):103-7. doi: 10.1016/j.brs.2008.09.009. Epub 2009 Feb 28. PMID 20633407
- [Background] Caumo W, Ruehlman LS, Karoly P, Sehn F, Vidor LP, Dall-Agnol L, Chassot M, Torres IL. Cross-cultural adaptation and validation of the profile of chronic pain: screen for a Brazilian population. Pain Med. 2013 Jan;14(1):52-61. doi: 10.1111/j.1526-4637.2012.01528.x. Epub 2012 Nov 21. PMID 23171145
- [Background] Sehn F, Chachamovich E, Vidor LP, Dall-Agnol L, de Souza IC, Torres IL, Fregni F, Caumo W. Cross-cultural adaptation and validation of the Brazilian Portuguese version of the pain catastrophizing scale. Pain Med. 2012 Nov;13(11):1425-35. doi: 10.1111/j.1526-4637.2012.01492.x. Epub 2012 Oct 4. PMID 23036076